CLINICAL TRIAL: NCT01011881
Title: Evaluation de la Mesure du Taux de la Procalcitonine Dans Les Liquides Pleuraux
Brief Title: Procalcitonin in Pleural Pleuritis
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI09-DR-DOUADI
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Pleuritis; Pleural Empyema
Keywords: pleuritis; empyema; procalcitonin
MeSH Terms: conditions — Pleurisy; Empyema, Pleural; Empyema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- patients with pleuritis
  Interventions: Other: pleural level of procalcitonin

INTERVENTIONS:
Other: pleural level of procalcitonin — no intervention

SUMMARY:
The purpose of this study is to determine pleural level of procalcitonin in differents situations of pleuritis.

DETAILED DESCRIPTION:
Determine pleural level of procalcitonin in pleuritis. Two periods First period evaluation in vitro study/ Determine adequat technique included type of samples tubes for adequat analysis.

Second periods : Patient with pleuritis . Empyema or not

ELIGIBILITY:
Inclusion Criteria:

* Pleuritis
* Hospitalisation

Exclusion Criteria:

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pleuritis
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2009-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France